CLINICAL TRIAL: NCT06543407
Title: Harm Reduction for Smokers With Mental Illness: RCT of E-cigarette Provision With or Without Behavioral Support to Boost Switching
Brief Title: Harm Reduction for Smokers With Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other); Fordham University (Other); Seven Counties Services (Unknown); Western Michigan University School of Medicine (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sarah Pratt, Associate Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02002328; R01DA057729-01A1 (NIH)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Dependence
Keywords: serious mental illness; harm reduction; e-cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Harm Reduction; Vaping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-cigarette provision only (Active Comparator): Participants randomized to this condition will receive a supply of NJOY Daily e-cigarettes for the first 8 weeks of the study.
  Interventions: Other: E-cig Provision Only
- SWITCH IT (Experimental): Participants randomized to this condition will receive a supply of e-cigarettes and behavioral support and coaching, protocolized intervention, SWITCH IT, for the first 8 weeks of the study.
  Interventions: Behavioral: SWITCH IT

INTERVENTIONS:
Behavioral: SWITCH IT — Behavioral support for switching, 7-10 sessions with SWITCH IT coach delivered during the first 8 weeks of the study. SWITCH IT participants will also have the opportunity to receive supported "field trips" to explore e-cigarette options based on availability, cost, and preferences during week 4 and week 6.
  Arms: SWITCH IT
Other: E-cig Provision Only — Provision of e-cigarettes (NJOY) based on combusible use for the first 8 weeks of the study.
  Arms: E-cigarette provision only

SUMMARY:
To compare the efficacy of e-cigarette (e-cig) provision with or without behavioral support (SWITCH IT) delivered via telehealth to reduce harm among smokers with MI who cannot quit smoking and are not ready to pursue cessation treatment, and to examine self-regulation (using e-cigs instead of cigarettes to cope with stress/distress and self-efficacy) as a potential mechanism for behavior change from SWITCH IT

ELIGIBILITY:
Diagnostic Criteria (must have one to be eligible):

* Schizophrenia
* Bipolar disorder
* Major Depressive Disorders
* Posttraumatic disorder
* Other anxiety disorders

Additional Inclusion Criteria:

* 21 years or older;
* English-speaking;
* Daily smoker (at least 10 cigarettes/day);
* At least one quit attempt in the past 5 years using evidence- based pharmacotherapy or behavioral cessation support;
* Not currently interested in quitting.

Exclusion Criteria:

* Currently residing in a nursing home;
* Current diagnosis of Asthma;
* Cognitive impairment (score <26 on the Telephone Interview for Cognitive Status (TICS);
* Current use of e-cigarettes (>once a week);
* Psychiatric instability (hospitalized in the past month);
* Current AND moderate to severe substance use disorder;
* Pregnant or planning to become pregnant;
* Use of any smoked products other than cigarettes;
* Current unstable medical illness making e-cigarette unsafe (e.g., recent heart attack, cancer);
* Participation in SWITCH IT pilot study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Urine NNAL | baseline to 8 weeks, 8 weeks to 26 weeeks
  urine levels of NNAL
Change in CO level | baseline to 8 weeks, 8 weeks to 26 weeks
  carbon monixide level less than 6
Change in self-reported cigarette use | baseline to 8 weeks 8 weeks to 16 weeks
  self-report of combustible cigarette use

CONTACTS AND LOCATIONS:
Overall Officials: Sarah I. Pratt, PhD, Principal Investigator — Dartmouth Health
Locations (2):
- United States (2):
  - Seven Counties Services, Louisville, Kentucky
  - The Providence Center, Providence, Rhode Island